CLINICAL TRIAL: NCT03678012
Title: Evaluation of Anti-biofilm Effects of Ferumoxytol (Feraheme) Using an in Situ Biofilm Demineralization Model
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 1802077294
Record Dates: First submitted 2018-09-07; First posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Ferrosoferric Oxide; Hydrogen Peroxide; Water

STUDY DESIGN:
Intervention Model Description: This will be a randomized, crossover, single blind in situ study with three test periods utilizing 16 subjects. The subjects in this study are lower partial denture wearers who have already had a study partial denture made for them as a part of a partial denture panel under 14-I-098 (IRB # 1407637739) or who will wear their own lower partial denture which was previously approved as part of the panel. The study partial dentures or personal partial dentures can house the specimen holders in two hollowed out areas of the buccal surface of two posterior denture teeth. The subjects will wear the lower partial dentures with enamel specimens in place for three consecutive 14-day study periods.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The study dentist, specimen/sample analysis technicians and the statistician will be blinded to the product allocation of subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ferumoxytol/Hydrogen peroxide (Active Comparator): 1.5% Ferumoxytol / 3% Hydrogen Peroxide (H2O2) 1:1 ratio
  Interventions: Drug: Ferumoxytol/Hydrogen peroxide
- Hydrogen peroxide (Placebo Comparator): Sham Solution / 3% Hydrogen Peroxide (H2O2) 1:1 ratio
  Interventions: Drug: Hydrogen Peroxide
- Water (Sham Comparator): Sham solution (water; negative control)
  Interventions: Drug: Water

INTERVENTIONS:
Drug: Ferumoxytol/Hydrogen peroxide — 1.5% Ferumoxytol / 3% Hydrogen Peroxide (H2O2) 1:1 ratio. Each subject will use this product during one of three treatment periods in the crossover study design.
  Other Names: Feraheme
  Arms: Ferumoxytol/Hydrogen peroxide
Drug: Hydrogen Peroxide — Sham Solution / 3% Hydrogen Peroxide (H2O2) 1:1 ratio. Each subject will use this product during one of three treatment periods in the crossover study design.
  Arms: Hydrogen peroxide
Drug: Water — Sham solution (water; negative control). Each subject will use this product during one of three treatment periods in the crossover study design.
  Arms: Water

SUMMARY:
To evaluate the effects of a clinically approved and commercially available iron oxide formulation Ferumoxytol (Feraheme®) to control cariogenic biofilms and enamel demineralization. This study will be testing topical application of Ferumoxytol extra-orally using a standard in situ biofilm demineralization model.

DETAILED DESCRIPTION:
This will be a randomized, crossover, single blind in situ study with three test periods utilizing 16 subjects. The subjects in this study are lower partial denture wearers who have already had a study partial denture made for them as a part of a partial denture panel under 14-I-098 (IRB # 1407637739) or who will wear their own lower partial denture which was previously approved as part of the panel. The study partial dentures or personal partial dentures can house the specimen holders in two hollowed out areas of the buccal surface of two posterior denture teeth. The subjects will wear the lower partial dentures with enamel specimens in place for three consecutive 14-day study periods.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 to 85 years of age and in good general and oral health without any known allergies to commercial dental products;
2. Evidence of a personally signed and dated informed consent document indicating the subject has been informed of all pertinent aspects of the trial;
3. Willingness to use the assigned products according to instructions, availability for appointments and likelihood of completing the clinical trial;
4. Willing to adhere to the study requirements and restrictions;
5. Lower partial denture wearers who have a lower partial denture made for them as a part of a partial denture panel under study 14-I-098 (IRB # 1407637739) or who agree to wear their own pre-approved lower partial denture that can house both specimens on one side of their partial denture.

Exclusion Criteria:

Oral Examination Inclusion Criteria:

1. Normal salivary flow rate (stimulated and unstimulated flow of ≥ 0.8 mL/min and ≥ 0.2 mL/min, respectively) ascertained from the Screening visit;
2. Willing and capable of wearing the lower partial denture 24 hours a day for the three, two-week treatment periods. Note: for persons who would otherwise qualify but whose lower partial denture needs repair, the individual may be listed as "pending". Once the partial denture has been repaired and adjusted to fit adequately for the subject to wear the lower partial denture 24 hours a day, the subject may be considered "qualified", complete their minimum 4 to 5 days washout period (of their own fluoridated toothpaste use) and continue with visit 2 in the study;
3. Absence of significant oral soft tissue pathology and dental caries, based on the dentist's visual examination and at the discretion of the investigator. Note: for persons who would otherwise qualify but who present at screening with dental caries requiring treatment, the individual may be listed as "pending". If the subject completes the restorative work within an acceptable amount of time, the subject may be considered qualified, complete their minimum 4 to 5 day washout period (of their own fluoridated toothpaste use) and continue with visit 2 in the study; and
4. Adequate oral hygiene (i.e. brush teeth daily and exhibit no signs of oral neglect).

Exclusion Criteria: Subjects presenting with any of the following will not be included in the trial:

1. Are taking or have ever taken bisphosphonate drugs (i.e., Fosamax, Actonel and Boniva) for the treatment of osteoporosis;
2. Use of blood thinning medications that prohibit the safe conduct of a dental cleaning (*NOTE: Subjects who are taking blood thinners in which written verification is obtained from their physician indicating their PT/INR levels (anti-coagulation blood levels) are at an acceptable level to avoid serious complications, such as bleeding during dental cleanings, may be accepted into the study);
3. Suspected alcohol or substance abuse (e.g., amphetamines, benzodiazepines, cocaine, marijuana, opiates) in the past year;
4. Report allergy to products (Ferumoxytol or other drugs or specific ingredients) used in the study, a reported history of multiple drug allergies or known hypersensitivity to any iron products;
5. Scheduled for MRI for the head region within three months after study participation involving Ferumoxytol application;
6. Have a history of significant adverse effects following the use of oral hygiene products such as dentifrices and mouth rinses;
7. Use of antimicrobial agents/antibiotics whether prescribed or over-the-counter within two weeks prior to each treatment visit;
8. Presence of severe marginal gingivitis or moderate/advanced periodontitis based on the clinical examination and discretion of the dental examiner;
9. Subjects who during the study will receive dental treatment, which may affect their participation (i.e. oral prophylaxis). Emergency treatment will be allowed if necessary;
10. Those requiring antibiotic premedication prior to dental treatment;
11. Participation in a dental clinical trial involving oral care products within 30 days of randomization (Baseline Visit);
12. Self-reported pregnancy or lactation or intent to become pregnant during the study period;
13. Self-reported chewing tobacco user;
14. Subjects who were previously screened and ineligible or were randomized to receive investigational product;
15. Significant unstable or uncontrolled medical condition, which may interfere with a subject's participation in the study;
16. Subjects who are related to those persons involved directly or indirectly with the conduct of this study; and
17. Other severe, acute or chronic, medical or psychiatric condition(s) or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

If the subject reports taking medication, a history of allergy, and/or a chronic disease which in the opinion of the investigator will not affect the clinical parameter(s) being assessed in this study or the safety of the subject, the subject may be enrolled in the study and it will be noted on the Investigator's source document.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-16 (Actual)

PRIMARY OUTCOMES:
Biofilm Analyses-cell viability | 14 days
  The effect of the treatments will be analyzed in terms of biochemical and microbiological composition of the biofilm formed. Colony forming unit (CFU) will be used to quantify the number of viable cells in biofilms.
Biofilm Analysis-extracellular polysaccharides | 14 days
  Biofilm EPS amount (weight in milligram) will be determined using colorimetric assay.

SECONDARY OUTCOMES:
Assessment of Enamel Demineralization by Means of Surface Microhardness Test (SMH) | 14 days
  The surface microhardness (SMH, length in micrometer) test will be used to assess changes in the mineral status of enamel specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Koo, Ph.D, Principal Investigator — University of Pennsylvania; Domenick Zero, Ph.D, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Oral Health Research Institute, Indianapolis, Indiana
  - University of Pennsylvania, School of dental medicine, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
No plan to share

REFERENCES:
- [Background] Cormode DP, Gao L, Koo H. Emerging Biomedical Applications of Enzyme-Like Catalytic Nanomaterials. Trends Biotechnol. 2018 Jan;36(1):15-29. doi: 10.1016/j.tibtech.2017.09.006. Epub 2017 Oct 26. PMID 29102240
- [Background] Gao L, Liu Y, Kim D, Li Y, Hwang G, Naha PC, Cormode DP, Koo H. Nanocatalysts promote Streptococcus mutans biofilm matrix degradation and enhance bacterial killing to suppress dental caries in vivo. Biomaterials. 2016 Sep;101:272-84. doi: 10.1016/j.biomaterials.2016.05.051. Epub 2016 Jun 2. PMID 27294544